CLINICAL TRIAL: NCT04052854
Title: A Single-Arm, Expanded Access Study of Zanubrutinib (BGB3111) in Participants With B-cell Malignancies
Brief Title: A Single-Arm, Expanded Access Study of Zanubrutinib in Participants With B-cell Malignancies
Status: No longer available | Type: Expanded Access
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Other Study IDs: BGB-3111-216
Record Dates: First submitted 2019-08-08; First posted 2019-08-12 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Waldenström Macroglobulinemia
Keywords: WM; Treatment naive; Relapsed/refractory
MeSH Terms: conditions — Waldenstrom Macroglobulinemia; Recurrence | interventions — zanubrutinib

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Zanubrutinib — Zanubrutinib will be orally administered in participants with treatment naive or R/R WM
  Other Names: BGB-3111

SUMMARY:
This is a multicenter expanded access study of zanubrutinib monotherapy for participants with B-cell malignancies who are ineligible to enroll into any available zanubrutinib clinical trials

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically confirmed diagnosis of WM with R/R disease or treatment-naive and considered by their treating physician to be unsuitable for standard chemoimmunotherapy regimens
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
3. Absolute neutrophil count (ANC) ≥ 0.75 x 109/L, independent of growth factor support; and Platelet count ≥ 50 x 109/L, independent of growth factor support or transfusion within 7 days of study entry
4. Creatinine clearance of ≥ 30 mL/min
5. Aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) ≤ 3 x upper limit of normal (ULN)
6. Total bilirubin level ≤ 2 x ULN (unless documented Gilbert's syndrome)

Key Exclusion Criteria:

1. Prior exposure to a Bruton tyrosine kinase (BTK) inhibitor
2. Evidence of disease transformation at the time of study entry
3. Ongoing requirement for systemic corticosteroid other than systemic adrenal replacement therapy
4. Chemotherapy given with antineoplastic intent, targeted therapy, radiation therapy or antibody-based therapy within 4 weeks of the start of study drug
5. Ongoing toxicity of ≥ Grade 2 from prior anticancer therapy
6. Prior or concurrent active malignancy within the past 2 years
7. Clinically significant cardiovascular disease
8. Unable to swallow capsules or disease significantly affecting gastrointestinal function
9. Active fungal, bacterial and/or viral infection requiring systemic therapy
10. Known infection with HIV, or serologic status reflecting active viral hepatitis B (HBV) or viral hepatitis C (HCV) infection as follows
11. Pregnant or lactating women
12. History of stroke or intracranial hemorrhage within 180 days before first dose of study drug
13. History of severe bleeding disorder
14. Active central nervous system (CNS) involvement by WM and/or lymphoma

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Brachmann, Study Director — BeiGene
Locations (10):
- United States (10):
  - Eisenhower Desert Cardiology Center, Rancho Mirage, California
  - Sansum Clinic and Ridley Tree Cancer Center, Santa Barbara, California
  - Maryland Oncology Hematology, Pa, Columbia, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Morristown Medical Center, Morristown, New Jersey
  - Icahn School of Medicine At Mount Sinai, New York, New York
  - Clinical Research Alliance, Inc, Westbury, New York
  - Texas Oncology Austin Midtown, Round Rock, Texas
  - Texas Oncology Tyler Longview, Tyler, Texas